CLINICAL TRIAL: NCT01174108
Title: Allogeneic Hematopoietic Stem Cell Transplantation for Severe Aplastic Anemia and Other Bone Marrow Failure Syndromes Using G-CSF Mobilized CD34+ Selected Hematopoietic Precursor Cells Co-Infused With a Reduced Dose of Non-Mobilized Donor T-Cells
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100154; 10-H-0154
Record Dates: First submitted 2010-07-31; First posted 2010-08-03 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-23

CONDITIONS: Severe Aplastic Anemia; MDS (Myelodysplastic Syndrome)
Keywords: Myelodysplastic Syndrome (MDS); Severe Aplastic Anemia; Pure Red Cell Aplasia; Paroxysmal Nocturnal Hemoglobinuria (PNH); Miltenyi CD34 Reagent System
MeSH Terms: conditions — Anemia, Aplastic; Anemia, Refractory, with Excess of Blasts; Myelodysplastic Syndromes; Red-Cell Aplasia, Pure; Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 1 (Experimental): Target doses: CD34+ cells 8 x 106/kg; CD3+ cells 2 x 107/kg
  Interventions: Device: Miltenyi CD34 Reagent System; Other: Donor derived G-CSF mobilized PBC
- 2 (No Intervention): Donor

INTERVENTIONS:
Device: Miltenyi CD34 Reagent System — The CliniMACS CD34 Reagent System is a medical device that is used in vitro to select and enrich specific cell populations.
  Arms: 1
Other: Donor derived G-CSF mobilized PBC — Cell Therapy
  Arms: 1

SUMMARY:
Background:

* Stem cell transplants from related donors (allogenic stem cell transplants) can be used to treat individuals with certain kinds of severe blood diseases or cancers, such as severe anemia. Allogenic stem cell transplants encourage the growth of new bone marrow to replace that of the recipient. Because stem cell transplants can have serious complications, researchers are interested in developing new approaches to stem cell transplants that will reduce the likelihood of these complications.
* By reducing the number of white blood cells included in the blood taken during the stem cell collection process, and replacing them with a smaller amount of white blood cells collected prior to stem cell donation, the stem cell transplant may be less likely to cause severe complications for the recipient. Researchers are investigating whether altering the stem cell transplant donation procedure in this manner will improve the likelihood of a successful stem cell transplant with fewer complications.

Objectives:

- To evaluate a new method of stem cell transplantation that may reduce the possibly of severe side effects or transplant rejection in the recipient.

Eligibility:

* Recipient: Individuals between 4 and 80 years of age who have been diagnosed with a blood disease that can be treated with allogenic stem cell transplants.
* Donor: Individuals between 4 and 80 years of age who are related to the recipient and are eligible to donate blood. OR unrelated donors found through the National Marrow Donor Program.

Design:

* All participants will be screened with a physical examination and medical history.
* DONORS:
* Donors will undergo an initial apheresis procedure to donate white blood cells.
* After the initial donation, donors will receive injections of filgrastim to release bone marrow cells into the blood.
* After 5 days of filgrastim injections, donors will have apheresis again to donate stem cells that are present in the blood.
* RECIPIENTS:
* Recipients will provide an initial donation of white blood cells to be used for research purposes only.
* From 7 days before the stem cell transplant, participants will be admitted to the inpatient unit of the National Institutes of Health Clinical Center and will receive regular doses of cyclophosphamide, fludarabine, and anti-thymocyte globulin to suppress their immune system and prepare for the transplant.
* After the initial chemotherapy, participants will receive the donated white blood cells and stem cells as a single infusion.
* After the stem cell and white blood cell transplant, participants will have regular doses of cyclosporine and methotrexate to prevent rejection of the donor cells. Participants will have three doses of methotrexate within the week after the transplant, but will continue to take cyclosporine for up to 4 months after the transplant.
* Participants will remain in inpatient care for up to 1 month after the transplant, and will be followed with regular visits for up to 3 years with periodic visits thereafter to evaluate the success of the transplant and any side effects.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (aHSCT) can cure patients with a variety of bone marrow failure syndromes (BMFS) including severe aplastic anemia (SAA), paroxysmal nocturnal hemoglobinuria (PNH) or myelodysplastic syndrome (MDS) associated with cytopenias. Patients with BMFS have traditionally been transplanted with bone marrow (BM) as a stem cell source. Although chronic graft versus host disease (cGVHD) occurs less commonly with BM compared to filgrastim (G-CSF) mobilized peripheral blood stem cell (PBSC) transplants, BM allografts have lower CD34+ progenitor cell numbers, which increases the risk of graft rejection in heavily transfused BMFS patients to 15-20%. To overcome this risk, our group developed a novel transplant approach for patients at high risk for graft rejection that utilized cyclophosphamide, fludarabine and anti-thymocyte globulin (ATG) conditioning followed by infusion of a CD34+ cell rich, T-cell replete G-CSF mobilized PBSC allograft. Remarkably, in 56 consecutive BMFS patients who had multiple risk factors for graft rejection who underwent this transplant approach, graft rejection did not occur, with all patients achieving complete donor lymphohematopoietic chimerism. Unfortunately, recipients of G-CSF mobilized PBSC had a higher incidence of cGVHD than has historically been observed with BM transplantation (72% vs. 50% cumulative incidence of cGVHD at 1 year respectively). G-CSF mobilized PBSC transplants contained approximately a 20 fold higher dose of T-cells that had undergone a TH-2 type cytokine polarization, a factor which likely contributed to this high incidence of cGVHD. In this protocol, we attempt to prevent graft failure and to reduce the incidence of cGVHD by transplanting high numbers of CD34+ selected PBSC co-infused with a reduced dose of non-mobilized donor T-cells that have not undergone a TH-2 cytokine polarization.

Subjects with BMFS at high risk for graft rejection will undergo allogeneic stem cell transplantation from an HLA identical sibling or match unrelated donor using the identical conditioning regimen utilized in protocol 99- H-0050. Using the Miltenyi CliniMACs system, recipients will receive an allograft on day 0 containing donor CD34+ cells that have been positively selected and T-cell depleted following G-CSF mobilization (goal CD34+ cell dose of 5 x 106 CD34+ cells /kg recipient) combined with 2 x 107 cells/kg of non-mobilized CD3+ T-cells previously collected and cryopreserved from the same donor by apheresis prior to G-CSF mobilization.

Primary objective: To evaluate whether administering a CD34+ selected, T-cell depleted peripheral blood stem cell graft with a concomitant infusion of non-mobilized donor T-cells at a dose that matches the T-cell dose that is infused in historical bone marrow transplant cohorts will reduce the incidence of cGVHD at 1 year to that observed with a conventional bone marrow transplant (50%) without increasing the risk of graft failure. This trial design will allow the trial to stop early if it is unlikely that we have reduced the proportion of one year cGVHD to 50% or if the combined event rate for failed donor engraftment or treatment related mortality (TRM) at day 100 exceeds 20%.

The primary endpoint of this study will be cGVHD at day 365.

Secondary end points include transplant related mortality, engraftment, degree of donor-host chimerism, incidence of acute and chronic graft versus host disease (cGVHD), transplant related morbidity and overall survival. Health related quality of life will also be assessed as a secondary outcome measure pre-transplant, 30 and 100 days post transplant, and every 6 months until 5 years post transplant.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Recipient:

  * Patients diagnosed with one of the following hematologic diseases which are associated with reasonable longevity, shown to be curable by allogeneic BMT but where concern for a high procedural mortality with conventional BMT may delay or prevent such treatment:

    * 1) Paroxysmal nocturnal hemoglobinuria (PNH) associated with life-threatening thrombosis, and/or cytopenia, and/or transfusion dependence and/or recurrent and debilitating hemolytic crisis
    * 2) Severe aplastic anemia (SAA) or pure red cell aplasia (PRCA [acquired or congenital]) with bone marrow cellularity <30% (excluding lymphocytes) associated with RBC or platelet transfusion dependence and/or neutropenia (absolute neutrophil count <=1000 cells/uL or for patients receiving granulocyte transfusions, absolute neutrophil count <=1000 cells/ uL before beginning granulocyte transfusions). in newly diagnosed patients and/or in patients who have failed immunosuppressive therapy.
    * 3) Refractory anemia (RA) or RARS MDS patients who have associated transfusion dependence and/or neutropenia.
  * Ages 4 to 80 (both inclusive), and weight >15 kg
  * Availability of HLA identical or single HLA locus mismatched family donor or 10/10 matched unrelated donor at the allelic level (HLA alleles A, B, C, DR, and DQ).
  * 9/10 donors where all the HLA sequences have the same antigen/peptide binding domains in key exons to the patient. This can result in identical protein sequences between patient and donor. Allele mismatches in p and g groups can be considered acceptable due to the exact matching which exists in the binding domains.
  * Telomere Length Testing
  * Germline/Inherited gene panel in patients where a suspicion for a familial bone marrow failure syndrome (BMFS) exist, hTERC and hTERT, GATA2 mutation testing will be performed on protocol 04-H-0012 or performed elsewhere prior to enrolling on 04-H-0012.

EXCLUSION CRITERIA:

- Recipient: any of the following

* Major anticipated illness or organ failure incompatible with survival from PBSC transplant
* Diffusion capacity of carbon monoxide (DLCO) <40% predicted (patients under the age of 10 may be excluded from this criterion if they have difficulty performing the test correctly and thus are unable to have their DLCO assessed) using DL Adj and DL/VA/Adj.
* Left ventricular ejection fraction <40% (evaluated by ECHO)
* Serum creatinine greater than 2.5mg/dl or creatinine clearance less than 50 ml/min by 24 hr urine collection
* Serum bilirubin greater than 4 mg/dl, transaminases greater than 5 times the upper limit of normal
* Pregnant or lactating
* Fanconi s anemia (test to be performed at a CLIA-certified laboratory)
* ECOG performance status of 3 or more (See NIH Bone & Marrow Transplant Consortium Supportive Care Guidelines for HSCT Recipients or Institutional Guidelines for bone and marrow transplants)
* Other malignant diseases liable to relapse or progress within 5 years, with the exception of a separate hematologic malignancy where allogeneic stem cell transplant has been shown to be potentially curative.
* Presence of an active infection not adequately responding to appropriate therapy.
* Inability to comprehend the investigational nature of the study and provide informed consent. The procedure will be explained to subjects age 8 -17 years with formal consent being obtained from parents or legal guardian.

INCLUSION CRITERIA:

-Related Donor:

* Related donor deemed suitable and eligible, and willing to donate, per clinical evaluations who are additionally willing to donate blood samples for research. Related donors will be evaluated in accordance with existing Standard Policies and Procedures for determination of eligibility and suitability for clinical donation. Note that participation in this study is offered to all related donors, but study participation is not required for a donor to make a stem cell donation, so it is possible that not all related donors will enroll onto this study
* Age greater than or equal to 4 and less than or equal to 80 years old

EXCLUSION CRITERIA:

-Related Donor: None

INCLUSION CRITERIA & EXCLUSION CRITERIA: Unrelated Donor

- The NMDP unrelated donor inclusion criteria will be used as outlined in document (http://bethematch.org/WorkArea/DownloadAsset.aspx?id=1960). Donor eligibility will be completed per NMDP standards and in accordance with most recent and stringent FDA guidelines.

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-12-10 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint of this study is chronic GVHD by one year. | 1 year
  chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - University of Maryland, Baltimore (UMB), Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
Currently the protocol does not specify whether the IPD will be shared. The prospect of IPD sharing is currently under consideration by the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-H-0154.html